CLINICAL TRIAL: NCT03108144
Title: Personalized Patient Alerts and Care Pathways to Prompt Prevention Interventions for Combined Alcohol and Tobacco Users in Primary Care
Brief Title: Personalized Alerts and Care Pathways to Prompt Prevention Interventions for Alcohol and Tobacco Users in Primary Care
Acronym: COMBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Dr. Peter Selby, Director, Medical Education, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 035-2015
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Cancer
Keywords: smoking cessation; alcohol; primary care; screening; brief intervention; referral to treatment; cancer risk
MeSH Terms: conditions — Neoplasms; Smoking Cessation | interventions — Ethanol; Methods

STUDY DESIGN:
Intervention Model Description: Organizations will be randomly allocated in a 1:1 allocation ratio to Group A (Test) or Group B (Control) accounting for rurality, organization type, practice size and academic affiliation.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Group A (No Intervention): When a patient is identified as consuming alcohol above CCS guidelines (based on mandatory baseline questionnaire) the practitioner in Group A will not receive computer alerts but will still have access to the alcohol consumption data as part of the baseline assessment (Screening). Healthcare providers will have access to all the same resources available as the intervention clinic (Treatment as usual).
- Intervention - Group B (Experimental): When a patient is identified as consuming alcohol above CCS guidelines (based on mandatory baseline questionnaire) the practitioner in Group B will receive computer alerts (Screening). The alert will provide a 5 minute script (Brief Intervention) for the health care providers to relay to patients and the ability to print or email a self-help resource to the patient each time the patient visits (Referral to Treatment).
  Interventions: Behavioral: Brief alcohol intervention

INTERVENTIONS:
Behavioral: Brief alcohol intervention — The intervention is a clinical decision support system (CDSS) that provides a computerized prompt in the clinic's online portal. The CDSS prompts a practitioner to intervene when a patient is screening above recommended drinking guidelines. The prompt appears as an alert message, recommending intervention. The portal suggests scripted brief intervention language, designed based on the College of Family Physicians of Canada and Canadian Centre on Substance Abuse's resource on conducting evidence-based Screening, Brief Intervention, and Referral to Treatment (SBIRT) guidelines.
  Arms: Intervention - Group B

SUMMARY:
Tobacco and alcohol use present multiplicative risk for aerodigestive cancers. Reducing alcohol consumption improves smoking cessation outcomes and reduces cancer risk. Risky alcohol consumption and smoking are often treated separately despite concurrent treatment potentially leading to better outcomes for each. However, no rapidly scalable program exists for combined interventions in primary care clinics spread across wide geographic areas. This cluster randomized trial aims to report on the effects of a novel clinical decision support system (CDSS) on intervention rates by primary care practitioners addressing risky alcohol use in a smoking cessation program.

The investigators will be implementing a clinical decision support system (CDSS) in 221 primary care sites participating in the Smoking Treatment for Ontario Patients (STOP) program across Ontario, Canada. Sites will be blindly allocated to one of two clinical decision support systems guiding practitioners to provide a risky alcohol use intervention to smokers attempting to quit using nicotine replacement therapy (NRT). Risky alcohol use is defined as drinking above the Canadian Cancer Society's low-risk drinking guidelines. Primary analysis will measure the proportion of risky drinkers offered an alcohol intervention in each CDSS arm at baseline. Patients will be contacted by phone or email to track smoking cessation and alcohol consumption rates at 6- and 12-month follow up.

Upon completion of the trial, the effect of different clinical decision support systems on practitioner behavior, and on client tobacco and alcohol use, will be discussed. If the CDSS successfully promotes SBIRT for risky alcohol use in a primary care setting and/or improves patient-level outcomes, including smoking cessation rates and alcohol use reduction, this tool can be used as a model for other web-based behavior change interventions integrated into primary care practice.

DETAILED DESCRIPTION:
Background: Primary care providers work in busy settings responding to a variety of acute and chronic problems. Implementing even brief evidence-based interventions for cancer risk behaviors, such as tobacco smoking and excess alcohol consumption, is sub-optimal due to time and knowledge constraints. These behaviors cluster in the same person and confer a multiplicative, positively associated risk for aero-digestive cancers but are often addressed separately, if at all, despite alcohol consumption undermining smoking cessation. Processes that reduce time and effort and yet increase practitioner effectiveness show promise to increase adoption of such practices. Computerized clinical decision support systems (CDSS) within practices allow for prompt procedural knowledge for practitioners, simplifies the decision-making process, and provides recommendations for patient care.

The initiation of the STOP Program (Smoking Treatment for Ontario Patients - an Ontario-wide initiative providing smoking cessation to eligible smokers who wish to quit), has demonstrated that such a system allows for rapid adoption of smoking cessation interventions in primary care with 189 sites (80% of eligible sites) in Ontario treating 40,000 smokers in 2 years. Approximately 36% consume alcohol above Canadian Cancer Society (CCS) guidelines (less than one drink per day for women; less then two drinks per day for men; no engagement in binge drinking) and those that do have a lower quit rate.

A combined alcohol and tobacco intervention delivered systematically using such a platform has never been studied before, which constitutes a missed opportunity to simultaneously address two closely related risk factors for cancer. Thus, implementation of a CDSS within the daily clinical workflow is a novel concept for cancer prevention with high potential to address the lack of brief interventions by health care providers.

Objective: Assess the effectiveness of a CDSS to increase the rates of brief alcohol intervention by healthcare providers and to reduce alcohol consumption in adult smokers making a quit attempt.

Methodology: Organizations from the STOP Program will be randomly allocated (1:1) to Group A or Group B.

Patient Population: Adult consenting smokers of the STOP Program identified as drinking above the sex-specific cut off at baseline will be eligible for the intervention.

Intervention: Half the sites will have a computer prompt built into STOP's data collection system, which will appear for any participant identified as drinking above the sex-specific cut off at baseline (Group A). The reminder will provide the practitioners with a five minute script advising their patient to reduce alcohol consumption to increase their chances of quitting smoking, and will be prompted to provide a self-help booklet to reduce alcohol intake. Sites without the prompt (Group B) will not receive reminders but will have access to the same resources.

ELIGIBILITY:
Inclusion Criteria:

* Participating clinics must be Family Health Team, Community Health Centre, or Nurse Practitioner-Led Clinic (primary care clinics) participating in the Smoking Treatment for Ontario Patients (STOP) program
* Clinic must use online portal to complete STOP questionnaires, in English, in real-time with patient

Exclusion Criteria:

* Non-primary care clinics participating in STOP program
* Clinics who conduct STOP questionnaires exclusively on paper, or in French, or not in real-time with patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15222 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Intervention offer by practitioner | Approximately 10 minutes during 1-hour appointment between practitioner and patient
  The study's primary outcome is the proportion of health practitioners who offer the brief alcohol intervention (with educational resource) to eligible patients.

SECONDARY OUTCOMES:
Intervention delivery by practitioner | Approximately 10 minutes during 1-hour appointment between practitioner and patient
  The study's secondary outcome is the proportion of health practitioners who deliver the brief alcohol intervention (with educational resource) to eligible patients (patient accepts practitioner's offer of intervention).
Smoking cessation and non-risky drinking | 6-month follow-up
  The study's tertiary outcome is the proportion of eligible participants who report being abstinent from smoking and meet CCS alcohol guidelines at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Selby, MBBS CCFP FCFP MHSc DipABAM, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minian N, Noormohamed A, Lingam M, Zawertailo L, Le Foll B, Rehm J, Giesbrecht N, Samokhvalov AV, Baliunas D, Selby P. Integrating a brief alcohol intervention with tobacco addiction treatment in primary care: qualitative study of health care practitioner perceptions. Addict Sci Clin Pract. 2021 Mar 16;16(1):17. doi: 10.1186/s13722-021-00225-x. PMID 33726843
- [Derived] Minian N, Baliunas D, Noormohamed A, Zawertailo L, Giesbrecht N, Hendershot CS, Le Foll B, Rehm J, Samokhvalov AV, Selby PL. The effect of a clinical decision support system on prompting an intervention for risky alcohol use in a primary care smoking cessation program: a cluster randomized trial. Implement Sci. 2019 Aug 23;14(1):85. doi: 10.1186/s13012-019-0935-x. PMID 31443663
- [Derived] Minian N, Noormohamed A, Zawertailo L, Baliunas D, Giesbrecht N, Le Foll B, Rehm J, Samokhvalov A, Selby PL. A method for co-creation of an evidence-based patient workbook to address alcohol use when quitting smoking in primary care: a case study. Res Involv Engagem. 2018 Feb 5;4:4. doi: 10.1186/s40900-018-0086-2. eCollection 2018. PMID 29445521
- [Derived] Minian N, Baliunas D, Zawertailo L, Noormohamed A, Giesbrecht N, Hendershot CS, Le Foll B, Rehm J, Samokhvalov A, Selby PL. Combining alcohol interventions with tobacco addictions treatment in primary care-the COMBAT study: a pragmatic cluster randomized trial. Implement Sci. 2017 May 18;12(1):65. doi: 10.1186/s13012-017-0595-7. PMID 28521782